CLINICAL TRIAL: NCT01720602
Title: A Pilot Study of Vorinostat to Restore Sensitivity to Aromatase Inhibitor Therapy Part B
Brief Title: Vorinostat in Treating Patients With Stage IV Breast Cancer Receiving Hormone Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7841; NCI-2012-02004 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Vorinostat; Anastrozole; Letrozole; exemestane; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vorinostat, AI therapy) (Experimental): Patients receive vorinostat PO 5 days a week for 3 weeks. Patients also receive AI therapy comprising either anastrozole PO daily, letrozole PO daily, or exemestane PO daily for 4 weeks. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: anastrozole; Drug: letrozole; Drug: exemestane; Procedure: positron emission tomography; Radiation: F-18 16 alpha-fluoroestradiol; Radiation: fludeoxyglucose F 18; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: anastrozole — Given PO
  Other Names: ANAS; Arimidex; ICI-D1033
Drug: letrozole — Given PO
  Other Names: CGS 20267; Femara; LTZ
Drug: exemestane — Given PO
  Other Names: Aromasin; FCE-24304; PNU 155971
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Radiation: F-18 16 alpha-fluoroestradiol — Correlative studies
  Other Names: F-18 FES; fluorine-18 16 alpha-fluoroestradiol
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies vorinostat in treating patients with stage IV breast cancer receiving hormone therapy. Vorinostat may help hormone therapy work better by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the rate of clinical benefit (objective response plus stable disease) for patients treated with 28-day cycles of vorinostat (first 5 consecutive days each week for day 1-21) concurrent with daily aromatase inhibitor (AI) therapy (all 28 days).

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of vorinostat and AI combination therapy in patients with metastatic breast cancer.

II. Assess the change in estrogen receptor (ER) expression, measured as the change in F-18 16 alpha-fluoroestradiol (FES) standardized uptake value (SUV) using FES positron emission tomography (PET) completed per protocol 7184 after two weeks of vorinostat and AI therapy and after 8 weeks of therapy.

III. Assess tumor metabolic response, measured as the change in fludeoxyglucose F 18 (FDG) SUV using FDG PET completed per protocol 7184 after two weeks of vorinostat and AI therapy and after 8 weeks of therapy.

IV. Assess the change in hormone levels (estradiol, estrone, follicle-stimulating hormone [FSH], sex binding globulin, testosterone, and free testosterone) after 8 weeks of therapy.

V. Assess the change in ER, progesterone receptor (PR), human epidermal growth factor receptor 2 (HER2), androgen receptor (AR), epidermal growth factor receptor (EGFR), vascular endothelial growth factor (VEGF) tumor expression after two weeks of vorinostat and AI therapy in patients that consent to optional tissue biopsy procedure.

VI. Assess the time to progression and the overall survival of patients treated with 28-day cycles of vorinostat (first 5 consecutive days each week for day 1-21) concurrent with daily AI therapy (all 28 days).

OUTLINE:

Patients receive vorinostat orally (PO) 5 days a week for 3 weeks. Patients also receive AI therapy comprising either anastrozole PO daily, letrozole PO daily, or exemestane PO daily for 4 weeks. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months until progression, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer
* Stage IV disease
* Patient has previously derived clinical benefit from endocrine therapy, but is no longer deriving benefit to endocrine therapy in the opinion of the treating investigator
* At least one site of measurable disease, as defined by the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Female patient is post menopausal as defined by one of the following; free from menses for >= 2 years, surgically sterilized, FSH and estradiol in post-menopausal range AND surgical absence of uterus OR chemotherapy induced amenorrhea lasting > 1 year OR currently on ovarian suppression
* Female patient of childbearing potential has a negative urine or serum (beta human chorionic gonadotropin [B-hCG]) pregnancy test within 14 days prior to receiving the first dose of vorinostat
* Male patient agrees to use two barrier methods of contraception or abstain from intercourse for the duration of the study
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 50,000/mcL
* Hemoglobin >= 9 g/dL
* Prothrombin time or international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) =< 1.2 times the ULN unless the patient is receiving therapeutic anticoagulation
* Potassium (K) levels normal limits
* Magnesium (Mg) levels normal limits
* Calculated creatinine clearance >= 30 mL/min

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent
* Patient has a life expectancy of at least 12 weeks in the opinion of the treating investigator
* Patient is willing to continue on same AI therapy
* Patient agrees to participate in imaging protocol 7184 and is separately consented

Exclusion Criteria:

* Patient has not derived clinical benefit from prior endocrine therapy
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug(s) other than the imaging protocol 7184
* Patient has received an ER blocking therapy (selective estrogen receptor modulating or downregulating selective estrogen receptor modulator [SERM] or selective estrogen receptor degrader [SERD] i.e. tamoxifen or fulvestrant) within the past 6 weeks
* Patient had prior treatment with an histone deacetylase (HDAC) inhibitor (e.g., romidepsin [Depsipeptide], NSC-630176, MS 275, LAQ-824, belinostat (PXD-101), LBH589, MGCD0103, CRA024781, etc); patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study; patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period
* Patient is on any systemic steroids that have not been stabilized to the equivalent of =< 10 mg/day prednisone during the 30 days prior to the start of the study drugs
* Patient has known hypersensitivity to the components of study drug or its analogs
* Patients with uncontrolled brain metastases
* New York Heart Association (NYHA) class III or IV congestive heart failure, myocardial infarction within the previous 6 months, QTc > 0.47 seconds, or uncontrolled arrhythmia
* Type I diabetes mellitus; patients with type II diabetes mellitus will be included as long as their glucose can be controlled to under 200 mg/dL
* Patient is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study
* Patient with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years or are considered by their physician to be at less than 30% risk of relapse
* Patients with known active viral hepatitis
* Patient has a history or current evidence of any condition, therapy, or laboratory (lab) abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vorinostat, AI Therapy)
Started | 15
Completed | 10
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Progressive disease on therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vorinostat, AI Therapy)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Benefit of Patients Receiving Vorinostat/AI Combination Therapy According to RECIST
Description: A 90% score (Wilson) confidence interval will be computed for the rate of clinical benefit.
  Clinical benefit according to Recist score is defined as: Stable Disease, Partial Remission or Complete Remission. Lack of clinical benefit is defined as Progressive Disease (increase in target lesion size by 20% or more).
Time Frame: 8 weeks
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Vorinostat, AI Therapy)
Number analyzed (Participants) | 10
percentage of patients | 60 [35 to 81]

2. Primary Outcome: Response Rate According to RECIST
Description: A 90% score (Wilson) confidence interval will be computed for the response rate.
  Clinical benefit according to Recist score is defined as: Stable Disease, Partial Remission or Complete Remission. Lack of clinical benefit is defined as Progressive Disease (increase in target lesion size by 20% or more).
Time Frame: 8 weeks
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Vorinostat, AI Therapy)
Number analyzed (Participants) | 10
percentage of patients | 60 [35 to 81]

3. Secondary Outcome: Duration of Response
Description: Duration of response will be summarized for responders.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Vorinostat, AI Therapy)
Number analyzed (Participants) | 6
weeks | 29.6 [24.9 to 91.4]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is assessed relative to the start of the study therapy. Progression can be determined by RECIST 1.1, elevated tumor markers, worsening clinical symptoms or new lesions identified by FDG-PET or bone scan.
Time Frame: From the time of start of study therapy to documented progression - up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Vorinostat, AI Therapy)
Number analyzed (Participants) | 15
months | 2 [0 to 21]

5. Secondary Outcome: Overall Survival
Description: Overall survival is assessed relative to the start of the study therapy to the date of death, from any cause.
Time Frame: From the time of start of study therapy to date of documented death
Population: OS includes one patient still alive 55 months after starting study therapy
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Vorinostat, AI Therapy)
Number analyzed (Participants) | 15
months | 19 [1 to 55]

ADVERSE EVENTS:
Arm/Group | Treatment (Vorinostat, AI Therapy)
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Vorinostat, AI Therapy) (N=15)
Liver failure (Hepatobiliary disorders) | 1 — Unrelated to the study treatment
Fever (Infections and infestations) | 1 — Unrelated to the study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Vorinostat, AI Therapy) (N=15)
decrease in glomerular filtration (Renal and urinary disorders) | 1 — grade 1 (CTCAE v3.0)
creatinine increase (Renal and urinary disorders) | 2 — grade 1-2 (CTCAE v3.0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 — grade 2 (CTCAE v3.0)
vomiting (Gastrointestinal disorders) | 2 — grade 2 (CTCAE v3.0)
diarrhea (Gastrointestinal disorders) | 1 — grade 3 (CTCAE v3.0)
nausea (Gastrointestinal disorders) | 2 — grade 2 (CTCAE v3.0)
neutropenia (Blood and lymphatic system disorders) | 1 — grade 3 (CTCAE v3.0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 — grade 2 (CTCAE v3.0)
Rigors / chills (General disorders) | 1 — grade 2 (CTCAE v3.0)
Dizziness (Nervous system disorders) | 1 — grade 3 (CTCAE v3.0) The relationship to vorinostat was unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No